CLINICAL TRIAL: NCT07160686
Title: A Phase III, Multicentre, Double Blind, Placebo-Controlled, Randomised Clinical Trial of Apixaban THROMBOprophylaxiS TO Prevent Venous Thromboembolism in Ambulatory Lung Cancer Patients Undergoing Systemic Anticancer Treatment
Brief Title: Apixaban to Prevent Venous Thromboembolism in Ambulatory Lung Cancer Patients Undergoing Systemic Anticancer Treatment
Acronym: THROMBO-STOP
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RG_25-043; NIHR165646 (Other Grant/Funding Number: NIHR Health Technology Assessment (NIHR HTA))
Record Dates: First submitted 2025-07-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Thromboprophylaxis
MeSH Terms: interventions — apixaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor's clinical trial management team other than the trial statisticians
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apixaban (Experimental): apixaban 2.5 mg twice a day for 6 months
  Interventions: Drug: Apixaban
- Placebo (Placebo Comparator): apixaban matched placebo twice a day for 6 months
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Apixaban — apixaban 2.5mg twice a day for 6 months
  Other Names: eliquis
  Arms: Apixaban
Other: Placebo — Placebo twice a day for 6 months
  Arms: Placebo

SUMMARY:
The aim of this trial is to find out if a tablet called apixaban can reduce blood clots in people with lung cancer having chemotherapy or similar treatments. Apixaban is a type of oral anticoagulant ("blood thinner") that makes the blood less sticky to prevent blood clots forming.

The trial is trying to find out if apixaban it can reduce blood clots in people with lung cancer.

Participants will receive the following treatment:

• Apixaban or placebo, 2.5mg taken by mouth twice a day for 6 months. This treatment will be taken in addition to any treatment that they are receiving to treat their lung cancer.

Participants will need to:

* Sign a consent form to enter the trial.
* Take the trial treatment as directed by the research team
* Complete a participant diary to record when they took the trial treatment
* Complete the Quality of Life and Health resource use questionnaires.
* Female participants of childbearing potential must use adequate contraception during the trial and for at least 2 days after trial treatment has finished.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is common in lung cancer and results in worse quality of life, increased healthcare costs, increased morbidity, and mortality. VTE is also increased in lung cancer patients undergoing systemic anticancer therapy (SACT). VTE can be reduced using anticoagulation as thromboprophylaxis, but this is not the current standard of care for outpatients having SACT. The subcutaneous anticoagulant low molecular weight heparin can reduce VTE in lung cancer but can be inconvenient to take. Apixaban is a type of direct oral anticoagulant (DOAC) taken in tablet form and not requiring regular blood monitoring, which have a good safety profile and are licensed for other medical conditions. Whilst anticoagulants have been used for thromboprophylaxis in patients with cancer, the role of DOACs in ambulatory lung cancer patients is unanswered by the existing literature.

THROMBO-STOP is a multicentre, double blind, placebo-controlled, parallel group, two arm, phase 3 randomised clinical trial testing the efficacy of Apixaban to reduce VTE in ambulatory lung cancer patients undergoing SACT. There will be a process evaluation, acceptability study and economic evaluation. For this superiority trial, 1456 patients (728 per group) are required to have a 90% power of detecting, as significant with an alpha of 0.05 (two-sided), a decrease in the rate of VTE from 8.6% in the control group (placebo) to 4% in the intervention group (apixaban), assuming a 20% drop-out rate. The planned recruitment of 1456 patients would involve 34 sites.

THROMBO-STOP patients will be recruited over a 36-month period which includes a 12-month internal pilot among a projected 40% of sites.

Data from these elements inform our stop/go criteria. The pilot aims to i) assess recruitment rate and exclusions ii) to assess VTE event rate iii) to assess progression criteria.

The overall study time will be 60 months accounting for trial set up and analysis.

Participants will be recruited to the trial from NHS UK sites.

Randomisation will be via a secure online system (staffed telephone back-up during office hours) based at CRCTU, allocating participants in a 1:1 ratio to either apixaban 2.5mg BD or placebo. A minimisation algorithm will be used within the system to ensure balance in the intervention allocations over the following variables: age (<70 or ≥70 ), sex (male or female) and cancer stage (III or IV). To avoid the possibility of the intervention allocation becoming predictable, a random element will be included in the algorithm.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 16 years
* Newly diagnosed locally advanced or metastatic primary lung cancer (histologically/ cytologically confirmed) or disease progression after complete or partial remission commencing a new course of SACT alone or as CRT
* Ambulatory (receiving outpatient SACT)

Exclusion criteria

* Hypersensitivity to apixaban or to any of the listed SmPC excipients
* Active clinically significant bleeding
* Lesion or condition considered a significant risk factor for major bleeding
* Hepatic disease associated with impaired synthetic function
* Platelet count < 50 x 109 /L
* Elevated liver enzymes ALT/AST > 2 x ULN or total bilirubin ≥ 1.5 x ULN
* Renal failure (creatinine clearance < 15ml/min)
* Weight < 40kg
* Estimated life expectancy < 6 months
* Continuous anticoagulation (e.g., unfractionated heparin, low molecular weight heparins, heparin derivatives and oral anticoagulants) for other medical conditions
* The usage of medications contraindicated with apixaban
* Pregnancy
* Breast feeding
* Judgement by the Investigator that the participant is unsuitable to participate in the trial and the participant is unlikely to comply with trial procedures, restrictions and requirements
* Inability to consent
* Receiving SACT for potentially resectable / resectable lung cancer as part of neo-adjuvant or adjuvant treatment
* SACT with significant potential DDI with apixaban (section 7.2.3)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 1456 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
18.3.1.1 Objectively confirmed VTE | 6 months
  Difference between a composite of objectively confirmed VTE and VTE-related death in participants with lung cancer, commencing SACT or CRT, when treated with 6 months of apixaban vs. placebo.

SECONDARY OUTCOMES:
Objectively confirmed VTE including all cause death | 6 months
  Composite of:
  i. New proximal or distal DVT (symptomatic or incidental) of upper or lower limbs, iliac veins, inferior/superior vena cava or central venous catheter related thrombosis ii. Non-fatal PE (symptomatic or incidental) iii. Death from any cause
Bleeding outcomes | 6 months
  * Major bleeding
  * Clinically relevant bleeding:
  Defined as the rate of participants experiencing at least one major bleeding and/or a clinically relevant non-major bleeding (CRNMB)
Net clinical benefit | 6 months
  Net clinical benefit (NCB) combines the primary efficacy outcome and major bleeding or clinically relevant bleeding. NCB is defined as: [the rate of VTE prevented by apixaban] minus [the rate of major or clinically relevant bleeding induced by apixaban].
  NCB= (VTE_control-VTE_apixaban ) - (Weighting × (Bleed_apixaban-Bleed_control )) VTE; the rate of objectively confirmed VTE or VTE related deaths (as defined for our primary outcome) Bleed; the rate of major bleeding or clinically relevant bleeding (as defined above).
  A default weighting factor of 1.0 will be used to represent an equal clinical weighting between the prevention of VTE by apixaban and the induction of major bleeding by apixaban, however supplementary analyses may be performed with a different weighting.
Proximal or distal DVT (symptomatic or incidental) | 6 months
  The rate of proximal or distal DVT will be collected and the Odds Ratio of apixaban vs placebo will be reported.
Other rates of thrombosis | 6 months
  The following thrombosis events will be investigated:
  * Arterial thromboembolism
  * Visceral thromboembolism
Survival outcomes | 6 months
  * VTE-related death
  * All cause death
  * Vascular death
EQ-5D-5L questionnaire | 6 months
  Questionnaires will be collected and the five subscale scores will be transformed to the summary index value using the value set(s) appropriate for the countries the trial opens in. Index values range from -0.285 and 1.00, with a higher score indicates a better quality of life. Median index values (along with subscale scores) will then be reported for apixaban and placebo groups, along with minimal important differences.
Time to VTE | 6 months
  VTE events (objectively confirmed VTE or VTE-related deaths) will be presented as a time to event outcome (time to VTE).
Non-fatal PE | 6 months
  The rate of non-fatal PEs will be collected and the Odds Ratio of apixaban vs placebo will be reported.
VTE-related death | 6 months
  Time to VTE-related death will be collected and the Hazard Ratio of apixaban vs. placebo will be reported.
Global EORTC QLQ-C30 questionnaire | 6 months
  Questionnaires will be collected and the mean global health status /QoL scale will be reported. This scale ranges from 0-100 with a higher score indicating a higher quality of life. Median health status/QoL (along with subscale scores) values will then be reported for apixaban and placebo groups, along with minimal important differences.
Lung cancer QLQ-LC29 questionnaire | 6 months
  Questionnaires will be collected and subscales will be calculated and reported. All subscales range from 0-100, with a higher score indicating a higher quality of life. Median values will then be reported for apixaban and placebo groups, along with minimal important differences

CONTACTS AND LOCATIONS:
Overall Officials: Michael Newnham, MBChB, MSc, MRCP, PhD, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available after the end of the study.
Supporting Information: Study Protocol
Time Frame: IPD and supporting information will be available within 12 months of the primary publication.
Access Criteria: Data anonymised in compliance with the Information Commissioners Office requirements, using a procedure based on guidelines from the Medical Research Council (MRC) Methodology Hubs and Information Commissioners Office, will be available for sharing with researchers outside of the trials team within 12 months of the primary publication.
URL: https://www.birmingham.ac.uk/research/centres-institutes/cancer-research-uk-clinical-trials-unit/data-sharing-policy